CLINICAL TRIAL: NCT05477368
Title: Examining the Feasibility of Prolonged Ketone Supplement Drink Consumption in Adults With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: H22-00644
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Diabetes; Hyperglycemia; Ketosis
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Ketosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exogenous Ketone Supplement (Experimental): Participants will be instructed to consume a total of 711 mL of the exogenous ketone supplement drink (for a total of 30 g of beta-hydroxybutyrate) per day (3 doses at 237 mL containing 10 g of beta-hydroxybutyrate each) for a period of 90 days.
  Interventions: Dietary Supplement: D-β-hydroxybutyric acid with R-1,3-butanediol
- Inert placebo (Placebo Comparator): Participants will be instructed to consume an equivalent volume (711 mL) of taste- and volume-matched placebo per day (3 doses at 237 mL) for 90 days.
  Interventions: Other: Inert placebo

INTERVENTIONS:
Dietary Supplement: D-β-hydroxybutyric acid with R-1,3-butanediol — Pre-intervention (baseline) and post-intervention measurements will be obtained before and after the 90-day period respectively.
  Arms: Exogenous Ketone Supplement
Other: Inert placebo — Pre-intervention (baseline) and post-intervention measurements will be obtained before and after the 90-day period respectively.
  Arms: Inert placebo

SUMMARY:
Ketones are a source of energy and signaling molecule that are produced by the body when not consuming any food or consistently eating a low-carbohydrate "keto" diet. Blood ketones can be used as a source of energy by the body, but they may also act as signals that impact how different cells in the body function.

Recently, ketone supplements have been developed that can be consumed as a drink. These supplements can raise blood ketones without having to fast or eat a "keto" diet. Previous studies have shown that these supplement drinks can lower blood sugar without having to make any other dietary changes. Drinking these ketone supplements may therefore be an effective strategy to improve blood sugar control and influence how cells function.

To find out if it is feasible for people with type 2 diabetes to drink these ketones supplements regularly over 90 days, we will compare between two groups in this study: one group that will be asked to drink ketone supplements, and one group that will be asked to drink a placebo supplement.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes by a physician at least 1 year prior
* stable use of glucose-lowering medications for at least three months
* must be able to read and understand English in order to complete the study questionnaires

Exclusion Criteria:

* competitively trained endurance athlete
* actively attempting to gain or lose weight
* having a history of mental illness or existing neurological disease
* having a history of cardiovascular events in the last two years, hypoglycemia, irritable bowel syndrome, or inflammatory bowel disease
* are currently taking SGLT2 inhibitors or insulin
* are using more than 2 classes of glucose-lowering medication
* currently following a ketogenic diet or regularly taking ketone supplements
* unable to commit to a 90-day trial
* being unable to follow remote guidance by internet or smartphone
* currently taking natural or over-the-counter supplements specifically designed to lower blood glucose (e.g., berberine, bitter melon)

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of conducting a randomized controlled trial (RCT) on the effects of consumption of a ketone supplement in adults with type 2 diabetes in free-living environment for 90 days: Recruitment rate of participants into the trial | Start of enrolment to completion of enrolment
  A recruitment rate of at least 4 participants per month (which will ensure the study is fully enrolled within a 1-year timeline) will be acceptable.
To determine the feasibility of conducting such an RCT: Compliance as measured by the self-reported volume of ketone supplement drink consumed | Across the 90-day intervention period (days 0 through 90)
  ≥ 67% of the drinks provided being consumed by participants as determined via self-report (i.e., an average of two out of three drinks per day being consumed) will be acceptable.
To determine the feasibility of conducting such an RCT: Retention as measured by the number of participants that complete the study | Across the 90-day intervention period (days 0 through 90)
  ≤ 30% of recruited participants dropping out of the study will be acceptable.

SECONDARY OUTCOMES:
Measures of glycemic control (HbA1c) | Day 0 (pre-intervention/baseline) and day 90 (post-intervention/follow-up)
  Glycemic control will be measured by assessing HbA1c in a clinical laboratory.
Measures of glycemic control (postprandial glucose area under the curve) | Days -5 through 9 (5 days of baseline and first 9 days of intervention period) and days 77 through 90 (last 2 weeks)
  Glycemic control will be measured by continuous glucose monitoring using the FreeStyle Libre 2 (Abbott) and quantified by assessing 2-hour postprandial hyperglycemia.
Measures of glycemic control (average daily glucose) | Days -5 through 9 (5 days of baseline and first 9 days of intervention period) and days 77 through 90 (last 2 weeks)
  Glycemic control will be measured by continuous glucose monitoring using the FreeStyle Libre 2 (Abbott) and quantified by assessing the average daily glucose.
Measures of glycemic control (glucose variability) | Days -5 through 9 (5 days of baseline and first 9 days of intervention period) and days 77 through 90 (last 2 weeks)
  Glycemic control will be measured by continuous glucose monitoring using the FreeStyle Libre 2 (Abbott) and quantified by assessing glucose variability.
Supplement acceptability | Days 1, 45, and 90
  Supplement acceptability will be assessed via questionnaire.
Gastrointestinal distress | Days 1, 45, and 90
  Gastrointestinal distress will be assessed via questionnaire.
Self-reported body weight | Day 0 (pre-intervention/baseline) and day 90 (post-intervention/follow-up)
  Self-reported body weight will be assessed by questionnaire.
Self-reported waist circumference | Day 0 (pre-intervention/baseline) and day 90 (post-intervention/follow-up)
  Self-reported waist circumference will be assessed by questionnaire (using study-provided measurement tape).
Self-reported energy consumption | Days 0 (pre-intervention/baseline), 45, and 90
  Self-reported energy consumption will be assessed via 24-hour dietary recalls.
Levels of perceived hunger | Days 0 (pre-intervention/baseline), 45, and 90
  Levels of perceived hunger will be assessed via questionnaire.
High-sensitivity c-reactive protein | Day 0 (pre-intervention/baseline) and day 90 (post-intervention/follow-up)
  High-sensitivity c-reactive protein will be measured in a clinical laboratory.
Hematology panel | Day 0 (pre-intervention/baseline) and day 90 (post-intervention/follow-up)
  Hematology panel will be measured in a clinical laboratory.
Liver enzymes (ALT, AST) | Day 0 (pre-intervention/baseline) and day 90 (post-intervention/follow-up)
  Liver enzymes (ALT, AST) will be measured in a clinical laboratory.
Lipid panel (triglycerides, total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, non-high density lipoprotein cholesterol, cholesterol/high-density lipoprotein cholesterol ratio) | Day 0 (pre-intervention/baseline) and day 90 (post-intervention/follow-up)
  Lipid panel will be measured in a clinical laboratory.
Levels of physical activity | Days 0 (pre-intervention/baseline), 45, and 90
  Levels of physical activity will be assessed via questionnaire.
Theory of planned behaviour | Days 0 (pre-intervention/baseline) and 45
  Theory of planned behaviour will be assessed via questionnaire.
Sleep quality | Days 0 (pre-intervention/baseline), 45, and 90
  Sleep quality will be assessed via questionnaire.
Cravings | Days 0 (pre-intervention/baseline), 45, and 90
  Cravings will be assessed via questionnaire.
Self-rated health | Days 0 (pre-intervention/baseline), 45, and 90
  Self-rated health and its impacts on daily life will be assessed via questionnaire.
Self-reported blood pressure (systolic and diastolic) | Days 0 (pre-intervention/baseline), 45, and 90
  Self-reported blood pressure (systolic and diastolic) will be assessed via questionnaire (via study-provided blood pressure monitors).

OTHER OUTCOMES:
Intervention acceptability | Across the 90-day intervention period (days 0 through 90)
  To evaluate the acceptability of the intervention and data collection procedures to participants, assessing the feasibility of implementing the intervention.
Viability of methods | Across the 90-day intervention period (days 0 through 90)
  To pilot methods for collecting outcome measures and ensure that our plans for recruitment, randomization, treatment, and follow-up are viable

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Little, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual patient data (de-identified) with researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The de-identified data and associated documents will be made available to researchers upon reasonable request for the duration that is required by the researchers.
Access Criteria: Researchers from accredited institutions will be granted access to the de-identified data and associated documents provided they can show that it will be used for a research-related purpose (e.g., meta-analysis).